CLINICAL TRIAL: NCT02366416
Title: Effects of Physical Exercise on Blood Glucose and Pain From the Musculoskeletal System in Patients With Type 2 Diabetes and Diabetes Related Complications
Brief Title: Effects of Physical Exercise on Blood Glucose and Pain From the Musculoskeletal System in Patients With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nordsjaellands Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-1-2014-122
Record Dates: First submitted 2015-02-05; First posted 2015-02-19 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Exercise, Physical
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Exercise training (Experimental): 12 weeks of one hour exercise training twice weekly
  Interventions: Behavioral: Exercise training

INTERVENTIONS:
Behavioral: Exercise training — Physical activity

SUMMARY:
The aim of this study is to investigate the effects og physical exercise on bloodglucose and pain from the musculoskeletal system in patients with type 2 diabetes.

The patients will be recruited to 12 weeks of exercise twice weekly. The outomes are long term bloodglucose (HbA1c) and pain reported in questionaires. In data analyses the patients will be stratified to patients with a high or a low degree of complications related to diabetes.

DETAILED DESCRIPTION:
Design: Uncontrolled intervention study Patients: Type 2 diabetes from Nordsjællands Hospital, Denmark Inclusion critera: adults, type 2 diabetes, not participating in an ungoing exercise program, able to conduct exercise training Exclusion criteria: unable to understand Danish, psychiatric disorder, dementia Intervention: two times one hour exercise training for 12 week. The training will be combined aerobic and resistance training supervised by physiotherapists Outcome: bloodglucose, pain (questionaire) Sample size: 80 participants

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Type 2 diabetes
* Must be able to perform physical exercise

Exclusion Criteria:

* Participation in structured exercise program within the past three months
* Dementia
* Unable to understand Danish language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Change of bloodglucose | Participants will be followed for a period of 12 weeks physical exercise
  HbA1c

SECONDARY OUTCOMES:
Change of musculoskeletal pain | Participants will be followed for a period of 12 weeks physical exercise
  Questionaire

CONTACTS AND LOCATIONS:
Overall Officials: Stig Moelsted, Phd, Principal Investigator — Nordsjaellands Hospital
Locations (1):
- Nordsjællands Hospital, Hillerød, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Molsted S, Tribler J, Snorgaard O. Musculoskeletal pain in patients with type 2 diabetes. Diabetes Res Clin Pract. 2012 May;96(2):135-40. doi: 10.1016/j.diabres.2011.12.022. Epub 2012 Jan 12. PMID 22244365
- [Background] Umpierre D, Ribeiro PA, Kramer CK, Leitao CB, Zucatti AT, Azevedo MJ, Gross JL, Ribeiro JP, Schaan BD. Physical activity advice only or structured exercise training and association with HbA1c levels in type 2 diabetes: a systematic review and meta-analysis. JAMA. 2011 May 4;305(17):1790-9. doi: 10.1001/jama.2011.576. PMID 21540423
- [Background] Thomas DE, Elliott EJ, Naughton GA. Exercise for type 2 diabetes mellitus. Cochrane Database Syst Rev. 2006 Jul 19;2006(3):CD002968. doi: 10.1002/14651858.CD002968.pub2. PMID 16855995
- [Background] Lebiedz-Odrobina D, Kay J. Rheumatic manifestations of diabetes mellitus. Rheum Dis Clin North Am. 2010 Nov;36(4):681-99. doi: 10.1016/j.rdc.2010.09.008. PMID 21092846